CLINICAL TRIAL: NCT00129402
Title: Efficacy, Safety, and Tolerability of Ezetimibe in Coadministration With Simvastatin in the Therapy of Adolescents With Heterozygous Familial Hypercholesterolemia
Brief Title: Effects of Ezetimibe With Simvastatin in the Therapy of Adolescents With HeFH (Study P02579)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P02579; EUDRACT NUMBER:2004-002627-40;; SCH 58235;; DOC ID 2526810
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Results first posted 2010-02-11 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: cholesterol; drugs; hypercholesterolemia; adolescent; randomized controlled trials
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Pooled subjects who received ezetimibe with simvastatin (Experimental): Pooled subjects who received ezetimibe 10 mg plus simvastatin 10 mg, simvastatin 20 mg, or simvastatin 40 mg
  Interventions: Drug: ezetimibe with simvastatin
- Pooled subjects who received simvastatin monotherapy (Active Comparator): Pooled subjects who received ezetimibe matching placebo plus simvastatin 10 mg, simvastatin 20 mg, or simvastatin 40 mg
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: ezetimibe with simvastatin — Ezetimibe 10 mg plus simvastatin 10 mg once a day for six weeks, or Ezetimibe 10 mg plus simvastatin 20 mg once a day for six weeks, or Ezetimibe 10 mg plus simvastatin 40 mg once a day for six weeks
  Arms: Pooled subjects who received ezetimibe with simvastatin
Drug: simvastatin — Ezetimibe matching placebo plus simvastatin 10 mg once a day for six weeks, or Ezetimibe matching placebo plus simvastatin 20 mg once a day for six weeks, or Ezetimibe matching placebo plus simvastatin 40 mg once a day for six weeks
  Arms: Pooled subjects who received simvastatin monotherapy

SUMMARY:
This is a randomized, double-blind, controlled, parallel-group, multicenter, Phase-3 study to evaluate the efficacy and safety of ezetimibe with simvastatin taken alone in subjects ages 10-17 years with Heterozygous Familial Hypercholesterolemia.

DETAILED DESCRIPTION:
This study consisted of 3 distinct periods. In Period 1, subjects received daily treatment for 6 weeks as part of either the ezetimibe with simvastatin group or part of the simvastatin monotherapy group. Subjects in the ezetimibe with simvastatin group received one of three treatments: coadministration of ezetimibe 10 mg/day plus simvastatin 10 mg/day, 20 mg/day, or 40 mg/day. Subjects in the simvastatin monotherapy group received one of three treatments: ezetimibe placebo plus simvastatin 10 mg/day, 20 mg/day, or 40 mg/day. The primary and key secondary efficacy analysis were based on the evaluations performed during Period 1 and were presented as data for subjects pooled from either the ezetimibe with simvastatin treatment groups compared with data for subjects pooled from the simvastatin monotherapy treatment groups.

In Period 2, subjects received ezetimibe 10 mg/day plus simvastatin 40 mg/day or ezetimibe placebo plus simvastatin 40 mg/day for 27 additional weeks maintaining the same treatment assignment (coadministration vs monotherapy) as in Period 1.

In Period 3, all subjects received ezetimibe 10 mg/day plus open-label simvastatin daily for 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent (ages 10 - 17 years) boys or girls weighing at least 88 lbs (40 kg).
* Subjects must have high cholesterol (low density lipoprotein cholesterol [LDL-C] more than 159 mg/dL or 4.1 mmol/L) and a family history of high cholesterol.

Exclusion Criteria:

* Subjects diagnosed with delayed puberty.
* Subjects who are sensitive to simvastatin and/or ezetimibe.
* Subjects who drink alcohol excessively or who have a history of alcohol or drug abuse within the past 2 years.
* Subjects who are known to be HIV positive, are undergoing LDL apheresis or plasma apheresis, or have had a partial ileal bypass.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

REFERENCES:
- [Derived] van der Graaf A, Cuffie-Jackson C, Vissers MN, Trip MD, Gagne C, Shi G, Veltri E, Avis HJ, Kastelein JJ. Efficacy and safety of coadministration of ezetimibe and simvastatin in adolescents with heterozygous familial hypercholesterolemia. J Am Coll Cardiol. 2008 Oct 21;52(17):1421-9. doi: 10.1016/j.jacc.2008.09.002. PMID 18940534

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe/Simvastatin 10/10: Subjects who received ezetimibe 10 mg plus simvastatin 10 mg once daily
- Ezetimibe/Simvastatin 10/20: Subjects who received ezetimibe 10 mg with simvastatin 10 mg once daily
- Ezetimibe/Simvastatin 10/40: Subjects who received ezetimibe 10 mg plus simvastatin 40 mg once daily
- Ezetimibe Matching Placebo/ Simvastatin 10: Subjects who received simvastatin monotherapy 10 mg once daily
- Ezetimibe Matching Placebo/ Simvastatin 20: Subjects who received simvastatin monotherapy 20 mg once daily
- Ezetimibe Matching Placebo/ Simvastatin 40: Subjects who received simvastatin monotherapy 40 mg once daily
- Long-term Experience Ezetimbe/Simvastatin: Subjects who received long-term coadministration of ezetimibe with simvastatin once daily
Period: Start Period1 to End Period1 (Week 1-6)
Arm/Group | Ezetimibe/Simvastatin 10/10 | Ezetimibe/Simvastatin 10/20 | Ezetimibe/Simvastatin 10/40 | Ezetimibe Matching Placebo/ Simvastatin 10 | Ezetimibe Matching Placebo/ Simvastatin 20 | Ezetimibe Matching Placebo/ Simvastatin 40 | Long-term Experience Ezetimbe/Simvastatin
Started | 43 | 40 | 43 | 40 | 40 | 42 | 0
Completed | 43 | 39 | 41 | 39 | 39 | 40 | 0
Not Completed | 0 | 1 | 2 | 1 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 0
Period: Start Period2 to End Period2 (Week 7-33)
Arm/Group | Ezetimibe/Simvastatin 10/10 | Ezetimibe/Simvastatin 10/20 | Ezetimibe/Simvastatin 10/40 | Ezetimibe Matching Placebo/ Simvastatin 10 | Ezetimibe Matching Placebo/ Simvastatin 20 | Ezetimibe Matching Placebo/ Simvastatin 40 | Long-term Experience Ezetimbe/Simvastatin
Started | 0 | 0 | 122 (# of subjects were combined from the 3 arms in Period 1 who received ezetimibe with simvastatin) | 0 | 0 | 118 (# of subjects were combined from the 3 arms in Period 1 who received simvastatin monotherapy) | 0
Completed | 0 | 0 | 114 (One subject who completed Period 1, did not enter Period 2, but entered and completed Period 3.) | 0 | 0 | 113 (One subject who completed Period 1, did not enter Period 2, but entered and completed Period 3.) | 0
Not Completed | 0 | 0 | 8 | 0 | 0 | 5 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Laboratory Adverse Event | 0 | 0 | 3 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 1 | 0
Period: Start Period3 to End Period3(Week 34-53)
Arm/Group | Ezetimibe/Simvastatin 10/10 | Ezetimibe/Simvastatin 10/20 | Ezetimibe/Simvastatin 10/40 | Ezetimibe Matching Placebo/ Simvastatin 10 | Ezetimibe Matching Placebo/ Simvastatin 20 | Ezetimibe Matching Placebo/ Simvastatin 40 | Long-term Experience Ezetimbe/Simvastatin
Started | 0 | 0 | 0 | 0 | 0 | 0 | 228 (In Period 3, all subjects from Period 1 and Period 2 were combined into one treatment group.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 222 (One subject who completed Period 1, did not enter Period 2, but entered and completed Period 3.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Subject moved | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pooled Subjects Who Received Simvastatin Monotherapy: Pooled subjects who received ezetimibe placebo plus simvastatin 10 mg, simvastatin 20 mg, or simvastatin 40 mg
- Total: Total of all reporting groups
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy | Total
Number analyzed (Participants) | 126 | 122 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (1.9) | 14.3 (1.8) | 14.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 73 | 69 | 142

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Least squares mean percent change from Baseline in LDL-C at the end of Step 1 (Week 6) in the pooled groups who received ezetimibe plus simvastatin compared with pooled groups who received simvastatin monotherapy
Time Frame: baseline to 6 weeks
Population: The analysis was performed on the intent to treat (ITT) population. Although 248 subjects received randomized treatment, two of the subjects did not have at least one baseline and at least one postbaseline lipid determination and thus could not be analyzed in the ITT population. Therefore, the actual ITT population consisted of 246 subjects.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy
Number analyzed (Participants) | 126 | 120
percent change | -49.45 (1.19) | -34.43 (1.22)
Statistical Analysis 1: Comparison: Pooled Subjects Who Received Ezetimibe With Simvastatin vs Pooled Subjects Who Received Simvastatin Monotherapy; Test type: Superiority or Other; p < 0.01, ANOVA

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Time Frame: baseline to 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Pooled Subjects Who Received Simvastatin Monotherapy: pooled subjects who received simvastatin 10 mg monotherapy, simvastatin 20 mg monotherapy, or simvastatin 40 mg monotherapy
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy
Number analyzed (Participants) | 126 | 120
percent change | -38.23 (.96) | -26.28 (.99)
Statistical Analysis 1: Comparison: Pooled Subjects Who Received Simvastatin Monotherapy; Test type: Superiority or Other; p < 0.01, ANOVA

3. Secondary Outcome: Percent Change From Baseline in Non High-density Lipoprotein Cholesterol (Non HDL-C)
Time Frame: baseline to 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy
Number analyzed (Participants) | 126 | 120
percent change | -46.84 (1.13) | -32.68 (1.16)
Statistical Analysis 1: Comparison: Pooled Subjects Who Received Ezetimibe With Simvastatin vs Pooled Subjects Who Received Simvastatin Monotherapy; Test type: Superiority or Other; p < 0.01, ANOVA

4. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG)
Time Frame: baseline to 6 weeks
Population: ITT
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy
Number analyzed (Participants) | 126 | 120
percent change | -16.56 (30.26) | -12.28 (31.49)
Statistical Analysis 1: Comparison: Pooled Subjects Who Received Ezetimibe With Simvastatin vs Pooled Subjects Who Received Simvastatin Monotherapy; Test type: Superiority or Other; p = .48, non-parametric model

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B)
Time Frame: baseline to 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy
Number analyzed (Participants) | 122 | 118
percent change | -38.92 (1.1) | -26.69 (1.11)
Statistical Analysis 1: Comparison: Pooled Subjects Who Received Ezetimibe With Simvastatin vs Pooled Subjects Who Received Simvastatin Monotherapy; Test type: Superiority or Other; p < 0.01, ANOVA

6. Secondary Outcome: Percent Change From Baseline in HDL-C
Time Frame: baseline to 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pooled Subjects Who Received Ezetimibe With Simvastatin | Pooled Subjects Who Received Simvastatin Monotherapy
Number analyzed (Participants) | 126 | 120
percent change | 6.58 (1.16) | 6.47 (1.19)
Statistical Analysis 1: Comparison: Pooled Subjects Who Received Ezetimibe With Simvastatin vs Pooled Subjects Who Received Simvastatin Monotherapy; Test type: Superiority or Other; p = .95, ANOVA

ADVERSE EVENTS:
Groups:
- Ezetimibe With Simvastatin: Column 1 provides the combined AE data collected for subjects in the ezetimibe with simvastatin treatment groups during Period 1 and Period 2
- Simvastatin Monotherapy: Column 2 provides the combined AE data collected for subjects in the simvastatin monotherapy treatment
  groups during Period 1 and Period 2.
- Long-term Coadministration of Ezetimibe With Simvastatin: Column 3 provides the combined AE data collected for
  all subjects that participated during Period 3. One subject who entered Period 3 did not receive study medication and was not included in the analysis.
Arm/Group | Ezetimibe With Simvastatin | Simvastatin Monotherapy | Long-term Coadministration of Ezetimibe With Simvastatin
Serious Adverse Events (participants affected / at risk) | 4/126 | 1/122 | 3/227
Other Adverse Events (participants affected / at risk) | 58/126 | 59/122 | 42/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe With Simvastatin (N=126) | Simvastatin Monotherapy (N=122) | Long-term Coadministration of Ezetimibe With Simvastatin (N=227)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe With Simvastatin (N=126) | Simvastatin Monotherapy (N=122) | Long-term Coadministration of Ezetimibe With Simvastatin (N=227)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (12) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 8 (9) | 12 (14) | 12 (12)
Nasopharyngitis (Infections and infestations) | 27 (30) | 27 (31) | 16 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 16 (25) | 16 (22) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9) | 5 (6)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less